CLINICAL TRIAL: NCT00002012
Title: Double-Blind, Randomized, Placebo-Controlled Study of Low Dose Oral Interferon Alfa-n3 (Human Leukocyte Derived) in ARC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Interferon Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 069A; 90-151ME
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Interferon Type I, Recombinant
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Interferon Alfa-n3

INTERVENTIONS:
Drug: Interferon alfa-n3

SUMMARY:
To conduct a parallel-group, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of an orally administered low dose interferon alfa-n3 as an immunomodulator in the treatment of mild to moderate symptomatic HIV+, AIDS-related complex (ARC) patients.

DETAILED DESCRIPTION:
The study has been extended to offer 52 weeks of maintenance therapy after the 10 weeks of the placebo controlled period are concluded successfully.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).

Patients must have:

* Diagnosis of AIDS related complex (ARC).
* Given written informed consent.
* Been receiving a dose of = or < 600 mg/day of zidovudine (AZT) at least 90 days prior to study entry IF they are currently taking AZT.

Prior Medication:

Allowed:

* Zidovudine (AZT) at a dose = or < 600 mg/day at least 90 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of AIDS-defining condition or evidence of AIDS dementia.
* Evidence of chronic hepatitis with severe liver dysfunction, or other active gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular or psychiatric disorder that would limit the subject's ability to complete the 12 weeks of the study period.

Concurrent Medication:

Excluded:

* Ketoconazole.
* Trimethoprim / sulfamethoxazole (TMP/SMX).
* Experimental medications.

Patients with the following are excluded:

* Absolute CD4 count of < 100 or > 350 cells/mm3.
* Any disease or disorder listed in Patient Exclusion Co-existing Conditions.
* Unlikely or unable to comply with the requirements of the protocol.
* Unwilling or unable to give informed consent.
* Development of antibodies to interferon during prior interferon therapy that occurred > 3 months prior to study entry.

Prior Medication:

Excluded within 45 days of study entry:

* Immunomodulators (e.g., BCG vaccine, isoprinosine).
* Chemotherapy.
* Steroids.
* Excluded within 3 months of study entry:
* Interferon therapy. Active IV drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Med Ctr, New York, New York, United States

REFERENCES:
- [Background] Hassett J, Mendelsohn L. Effect of low dose oral interferon alfa-n3 (IFN) in ARC. Int Conf AIDS. 1993 Jun 6-11;9(1):494 (abstract no PO-B28-2151)